CLINICAL TRIAL: NCT01879774
Title: Characterisation of Neuropsychological and Motoric Performance in Patients With Hyponatremia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, Principal Investigator, University of Cologne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 002
Record Dates: First submitted 2013-04-23; First posted 2013-06-18 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Hyponatremia
Keywords: Hyponatremia
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with hyponatremia (Other): Neuropsychological and motoric tests are conducted in patients with hyponatremia.
  Interventions: Other: Neuropsychological and motoric tests
- Patients with normal serum sodium (Other): Neuropsychological and motoric tests are conducted in patients with normal serum sodium.
  Interventions: Other: Neuropsychological and motoric tests

INTERVENTIONS:
Other: Neuropsychological and motoric tests — 1. Neuropsychological tests
     * Mini Mental Status Test
     * Dem-Tect
     * Rey-Osterrieth Complex Figure Test
     * Trailmaking Test
     * Beck Depression Inventory
     * d2-R (optional)
  2. Motoric tests
     * modified UPDRS (Unified Parkinson Disease Rating Scale) Part III
     * Timed-up-and-go Test
     * Halstead Fingertapping Test
     * AIMS (Abnormal involuntary movement scale)
  3. EEG (only in patients with hyponatremia)
  4. MRI (only in patients with hyponatremia)

SUMMARY:
The aim of this epidemiological study is to characterize the neuropsychological and motoric performance in patients with hyponatremia. Newer studies revealed an association between mild hyponatremia and unstable walking, frequency of falls and risk of a fracture, questioning the paradigm of an "asymptomatic" hyponatremia. Until now, there is no known detailed investigation and characterisation of the cognitive and motoric performance or limitation by this disorder. Therefore this study will investigate patients with hyponatremia on the basis of neuropsychological and neurological tests.

DETAILED DESCRIPTION:
Hyponatremia is the most common electrolyte disorder in outpatients and hospitalized patients. The prevalence of hospital-associated hyponatremia is estimated to be up to 40%. Especially mild to moderate hyponatremia (125-136 mmo/l) without apparent symptoms has seldomly been accurately assessed but rather seen as clinically irrelevant. Cognitive limitations, unstable gait and motoric disorders as well as depressive conditions were described in smaller studies and single case reports.

In terms of the question, if a therapeutic influence is also reasonable in slight symptomatic hyponatremia it is necessary to establish an accurate phenotyping of patients with hyponatremia, which quantifies the individual cognitive, motoric and psychological qualities.

Patients with hyponatremia will be examined on the basis of standardized neuropsychological and neurological tests. Following questions are to be answered with this study:

1. Which cognitive, motoric and psychological functions are impaired due to hyponatremia?
2. Is there a correlation between the extend of hyponatremia and the different test results?
3. Is there an intraindividual difference in test results during hyponatremia and normal sodium concentrations?

In addition to clinical testing, functional magnetic resonance imaging (fMRI) will be performed before and after therapy in up to 40 patients with hyponatremia. Functional magnetic resonance imaging (fMRI) is an imaging procedure in which local changes in cerebral oxygen concentration can be used to draw conclusions about brain activity. In connection with the current research project, an initial contribution is to be made in order to close the existing knowledge gap as to whether a functionally-image-morphologically tangible change in cerebral activity can also be depicted non-invasively by means of fMRI during hyponatremia or after its compensation. Another component of cerebral evaluation in this context is volumetry in fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or older
* Hyponatremia with serum sodium < 130 mmol/l
* Men and women with normal serum sodium > 130 mmol/l (control group)

Exclusion Criteria:

* traumatic cerebral injury, hemorrhagic and ischemic insult as cause of hyponatremia
* professional or private relationship between subject and the investigators, or dependance on the investigators
* Placement in an institution based on official orders
* Patients who are unable to give informed consent
* Patients with contraindication for MRI investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Assessment of Performance in individual tests | Change in individual tests at Baseline and at least 48 hours after first assessment

SECONDARY OUTCOMES:
Assessment of cerebral basal activity in fMRI during hyponatremia and after its compensation | Change in fMRI from baseline and at least 48 hours after first assessment

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Principal Investigator — University Hospital of Cologne
Locations (3):
- University of Cologne, Cologne, Germany
- Dipartimento di Scienze Biomediche, Sperimentali e Cliniche Mario Serio, Florence, Italy
- Hospital Universitario Clinico San Carlos, Madrid, Spain